CLINICAL TRIAL: NCT02567084
Title: A Prospective, Longitudinal Patient Study on CERAMENT™|BONE VOID FILLER in Benign Bone Tumors
Brief Title: Complete Twelve Month Bone Remodeling With a Bi-phasic Injectable Bone Substitute in Benign Bone Tumors
Acronym: BRBBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, M.D Maciej Goch, Principal Investigator, Poznan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POZNAN-UMS-JK1
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Bone Cyst
Keywords: Bone substitute; benign bone cyst; ceramic; remodelling
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CERAMENT™ |BONE VOID FILLER (Other): Intraoperativ application of medical device: CERAMENT™ |BONE VOID FILLER 5cc/10cc/18cc
  Interventions: Device: CERAMENT™ |BONE VOID FILLER

INTERVENTIONS:
Device: CERAMENT™ |BONE VOID FILLER — Implantation of bi-phasic ceramic bone substitute to provide bone generation and bone remodeling in patients with benign bone tumors.

SUMMARY:
The purpose of this study is to assess the ability a injectable bi-phasic ceramic bone substitute to provide bone generation and bone remodeling in patients with benign bone tumors.

DETAILED DESCRIPTION:
The aim of the study is to assess the usefulness of injectable bi-phasic ceramic bone substitute (CERAMENT™ |BONE VOID FILLER) in patients with benign bone tumors. The primary objectives is to:

1. Assess the ability of bi-phasic ceramic bone substitute to provide bone generation and bone remodeling in patients with benign bone tumors.
2. Assess the safety of bi-phasic ceramic bone substitute as measured by device complaint/Adverse Events monitoring and documentation of subsequent surgical procedure.
3. In the case of bone cysts assess the ability of bi-phasic ceramic bone substitute to transform into bone and possibly induce bone formation in regions of the cyst not filled with the product.

Benign bone tumors are often treated with intralesional curettage which creates a bone defect that can be filled with e.g. demineralized bone matrix, autologous bone, ceramic bone substitutes or polymethylmetacrylate cement.

Autograft has been considered the golden standard because it possesses all three of the essential elements required for an optimal bone graft, but is associated with morbidity at the donor site and is limited in supply. Allograft has been employed as a good alternative to autograft but the concern for potential disease transmission remains. Synthetic bone graft substitutes have been gaining popularity as viable alternatives for void and defect filling eliminating the concerns with autograft and allograft. These synthetic bone substitutes have invariably been based on calcium phosphate and/or calcium sulfate materials which are osteoconductive and facilitate bone remodeling, although side effects such as drainage and wound complications slow remodeling to bone or negligible bone generation have limited their use. Thus, new synthetic bone substitutes with described positive effects in vertebroplasty, osteotomy, and smaller trauma defects merit further investigation also in treatment of larger bone defects.

In a prospective series, patients with benign bone tumors were treated by minimal invasive intervention with a bi-phasic and injectable ceramic bone substitute (CERAMENT™ BONE VOID FILLER), composed of 60% weight synthetic calcium sulfate (CaS) and 40% weight hydroxyapatite (HA) powder was mixed with a water-soluble radio-contrast agent iohexol (180 mg/ml) to make the material radiopaque. The defects were treated by either mini-invasive surgery (solid tumors) or percutaneous injection (cysts) and followed clinically and radiologically for 12 months. CT scan was performed after 12 months to confirm bone remodeling of the bone substitute. All patients were allowed full weight bearing immediately after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital for surgical treatment of benign bone lesion requiring bone grafting.

Exclusion Criteria:

* Patient below 6 years of ageIrreversible coagulopathy or bleeding disorder. Note regarding reversible coagulopathies: Patients on coumarin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re-initiation of anticoagulants;
* A pre-existing calcium metabolism disorder (e.g. hypercalcemia).

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
bone remodeling according to Neer classification | 12 months after surgery
  Evaluate bone healing and remodeling at 12 month by X-ray and CT-scan using Modified Neer classification of radiological results.

SECONDARY OUTCOMES:
cyst and bone formation volume | 12 months after surgery
  Calculate the pre-operative volume of the cyst, document the volume of product placed into the cyst and the volume of bone formed at 12 months.
  In the case of bone cysts assess the ability of CERAMENT™ |BONE VOID FILLER to transform into bone and possibly induce bone formation in regions of the cyst not filled with the product.
adverse events | 12 months after surgery
  Assess the safety of CERAMENT™|BONE VOID FILLER as measured by number of any device complaint/Adverse Event and any subsequent surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kaczmarczyk, Prof.MD,PhD, Principal Investigator — Poznan Medical University

REFERENCES:
- [Background] Mik G, Arkader A, Manteghi A, Dormans JP. Results of a minimally invasive technique for treatment of unicameral bone cysts. Clin Orthop Relat Res. 2009 Nov;467(11):2949-54. doi: 10.1007/s11999-009-1008-2. Epub 2009 Aug 4. PMID 19653053
- [Background] Khan SN, Tomin E, Lane JM. Clinical applications of bone graft substitutes. Orthop Clin North Am. 2000 Jul;31(3):389-98. doi: 10.1016/s0030-5898(05)70158-9. PMID 10882465
- [Background] Myeroff C, Archdeacon M. Autogenous bone graft: donor sites and techniques. J Bone Joint Surg Am. 2011 Dec 7;93(23):2227-36. doi: 10.2106/JBJS.J.01513. PMID 22159859
- [Background] Hinsenkamp M, Muylle L, Eastlund T, Fehily D, Noel L, Strong DM. Adverse reactions and events related to musculoskeletal allografts: reviewed by the World Health Organisation Project NOTIFY. Int Orthop. 2012 Mar;36(3):633-41. doi: 10.1007/s00264-011-1391-7. Epub 2011 Nov 3. PMID 22048753
- [Background] Lee GH, Khoury JG, Bell JE, Buckwalter JA. Adverse reactions to OsteoSet bone graft substitute, the incidence in a consecutive series. Iowa Orthop J. 2002;22:35-8. PMID 12180608
- [Background] Ferguson JY, Dudareva M, Riley ND, Stubbs D, Atkins BL, McNally MA. The use of a biodegradable antibiotic-loaded calcium sulphate carrier containing tobramycin for the treatment of chronic osteomyelitis: a series of 195 cases. Bone Joint J. 2014 Jun;96-B(6):829-36. doi: 10.1302/0301-620X.96B6.32756. PMID 24891586
- [Background] Reppenhagen S, Reichert JC, Rackwitz L, Rudert M, Raab P, Daculsi G, Noth U. Biphasic bone substitute and fibrin sealant for treatment of benign bone tumours and tumour-like lesions. Int Orthop. 2012 Jan;36(1):139-48. doi: 10.1007/s00264-011-1282-y. Epub 2011 May 28. PMID 21626113
- [Background] Fillingham YA, Lenart BA, Gitelis S. Function after injection of benign bone lesions with a bioceramic. Clin Orthop Relat Res. 2012 Jul;470(7):2014-20. doi: 10.1007/s11999-012-2251-5. PMID 22290129
- [Background] Petruskevicius J, Nielsen S, Kaalund S, Knudsen PR, Overgaard S. No effect of Osteoset, a bone graft substitute, on bone healing in humans: a prospective randomized double-blind study. Acta Orthop Scand. 2002 Oct;73(5):575-8. doi: 10.1080/000164702321022875. PMID 12440503
- [Background] Hatten HP Jr, Voor MJ. Bone healing using a bi-phasic ceramic bone substitute demonstrated in human vertebroplasty and with histology in a rabbit cancellous bone defect model. Interv Neuroradiol. 2012 Mar;18(1):105-13. doi: 10.1177/159101991201800114. Epub 2012 Mar 16. PMID 22440608
- [Background] Masala S, Nano G, Marcia S, Muto M, Fucci FP, Simonetti G. Osteoporotic vertebral compression fracture augmentation by injectable partly resorbable ceramic bone substitute (Cerament|SPINESUPPORT): a prospective nonrandomized study. Neuroradiology. 2012 Nov;54(11):1245-51. doi: 10.1007/s00234-012-1016-x. Epub 2012 Mar 6. PMID 22391680
- [Background] Abramo A, Geijer M, Kopylov P, Tagil M. Osteotomy of distal radius fracture malunion using a fast remodeling bone substitute consisting of calcium sulphate and calcium phosphate. J Biomed Mater Res B Appl Biomater. 2010 Jan;92(1):281-6. doi: 10.1002/jbm.b.31524. PMID 19904822
- [Background] Nilsson M, Zheng MH, Tagil M. The composite of hydroxyapatite and calcium sulphate: a review of preclinical evaluation and clinical applications. Expert Rev Med Devices. 2013 Sep;10(5):675-84. doi: 10.1586/17434440.2013.827529. PMID 24053255
- [Background] Sung AD, Anderson ME, Zurakowski D, Hornicek FJ, Gebhardt MC. Unicameral bone cyst: a retrospective study of three surgical treatments. Clin Orthop Relat Res. 2008 Oct;466(10):2519-26. doi: 10.1007/s11999-008-0407-0. Epub 2008 Aug 5. PMID 18679761
- [Background] Cho HS, Seo SH, Park SH, Park JH, Shin DS, Park IH. Minimal invasive surgery for unicameral bone cyst using demineralized bone matrix: a case series. BMC Musculoskelet Disord. 2012 Jul 29;13:134. doi: 10.1186/1471-2474-13-134. PMID 22839754
- [Background] Campanacci M, Capanna R, Fabbri N, Bettelli G. Curettage of giant cell tumor of bone. Reconstruction with subchondral grafts and cement. Chir Organi Mov. 1990;75(1 Suppl):212-3. No abstract available. PMID 2249537
- [Background] Bickels J, Meller I, Shmookler BM, Malawer MM. The role and biology of cryosurgery in the treatment of bone tumors. A review. Acta Orthop Scand. 1999 Jun;70(3):308-15. doi: 10.3109/17453679908997814. PMID 10429612
- [Derived] Kaczmarczyk J, Sowinski P, Goch M, Katulska K. Complete twelve month bone remodeling with a bi-phasic injectable bone substitute in benign bone tumors: a prospective pilot study. BMC Musculoskelet Disord. 2015 Nov 26;16:369. doi: 10.1186/s12891-015-0828-3. PMID 26612576